CLINICAL TRIAL: NCT05052632
Title: Evaluating a New Gonadotoxic Risk Stratification System
Status: Withdrawn | Type: Observational
Why Stopped: Cancelled by PI
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3084
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: ovarian reserve
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study is to assess if there is an association between a newly described gonadotoxic risk stratification system and post-treatment ovarian reserve as determined by FSH and AMH.

DETAILED DESCRIPTION:
The Investigator will test the amount of agreement between the two ordinal variables using a kappa statistic at each time point in the first two years of follow up. The Investigator will perform ordinal logistic regression accounting for repeated measures data for participants who are not using contraception. The Investigator will assess participant characteristics to see if the Investigator need to adjust for other covariates including age, race, ethnicity and body mass index (BMI).

Since contraception can mask an elevated FSH surge from gonadal failure, the Investigator will perform a similar model for participants on contraception using AMH only.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ages 8 - 39 years of age
* Seen in CHCO or AMC outpatient clinics for any of the following reasons:

  * At risk for fertility problems (Z91.89)
  * Encounter for fertility preservation counseling (Z31.62)
  * Primary ovarian insufficiency
  * Premature ovarian failure/premature menopause
  * Diminished ovarian reserve
* At least 12 months post-completion of chemotherapy and/or radiation
* History of a fertility-threatening diagnosis receiving chemotherapy; radiation; or surgery to the reproductive organs for malignancy, including but not limited to:

  * Any type of cancer/malignancy
  * Rheumatoid arthritis
  * Systemic lupus erythematosus
  * Aplastic anemia
  * Fanconi anemia
  * Diamond-Blackfan syndrome
  * Hurler syndrome
  * Other autoimmune conditions

Exclusion Criteria:

* Disorders of sexual development (i.e., gonadal dysgenesis, Turner syndrome/mosaicism, etc.)
* History of bilateral oophorectomy
* Transgender patients not receiving chemotherapy; radiation; or surgery to the reproductive organs for malignancy
* Inability to consent/assent

Ages: 8 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — In this study the Investigator is looking at Ovarian reserve and only female population will be included.
Study Population: Study participants will be prepubertal (8-12 years) and post-pubertal (13-39) females seen at the University of Colorado Anschutz Pavilion and/or Children's Hospital Colorado who have received gonadotoxic chemotherapy; radiation; or surgical excision of a reproductive organ for malignancy. The study participants will be assessed based on whether they are pre- or post-pubertal and then further stratified by age < 25 years and > 25 years based on the expected age-related decline of AMH.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve | 2 year follow up
  The Investigator will evaluate if there is an association between ovarian reserve (defined using AMH and FSH) and the risk stratification system categories (minimally increased risk, significantly increased risk, and high level of increased risk). Specifically Ovarian reserve goes from normal ([FSH <10] AND [AMH >= 1.0]), Diminished ovarian reserve ([10 <=FSH < 25] or [ 0.5 <= AMH <1.0]), primary ovarian insufficiency ([25<= FSH] or [ 0.5 < AMH]). AMH: ng/ml, FSH: mIU/ml. Investigator will test the amount of agreement between the two ordinal variables using a kappa statistic at each time point in the first two years of follow-up. Investigator will perform ordinal logistic regression accounting for repeated measures for participants who are not using contraception. Investigator will access patient characteristics to see if Investigator need to adjust for other covariates including age, race, ethnicity, and body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Appiah, MD, Principal Investigator — University of Colorado, Denver